CLINICAL TRIAL: NCT00471380
Title: A Phase IV Study of Travoprost + Brinzolamide to Treat Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IT-04-04; EudraCT 200600362737
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; dorzolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crossover group ABB (Active Comparator): 3 period, 2 treatment cross-over model:
  Participants received Treatment A, which was concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.) for period 1 for 8 weeks. Then participants received Treatment B, which was fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.) for Period 2 (8 weeks) and Period 3 (8 weeks)
  Interventions: Drug: travoprost 0.004% and brinzolamide 1%; Drug: fixed combination of timolol 0.5% and dorzolamide 2% plus travoprost vehicle
- Crossover group BAA (Active Comparator): 3 period, 2 treatment cross-over model:
  Participants received Treatment B, which was fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.) for Period 1 (8 weeks). Then participants received Treatment A, which was concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.) for Period 2 (8 weeks) and Period 3 (8 weeks).
  Interventions: Drug: travoprost 0.004% and brinzolamide 1%; Drug: fixed combination of timolol 0.5% and dorzolamide 2% plus travoprost vehicle

INTERVENTIONS:
Drug: travoprost 0.004% and brinzolamide 1% — Group A = concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.)
Drug: fixed combination of timolol 0.5% and dorzolamide 2% plus travoprost vehicle — group B = fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.).

SUMMARY:
Double blind, crossover randomized, multicentric study to compare efficacy and tolerability of concomitant administration of travoprost and brinzolamide versus timolol-dorzolamide fixed combination in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of bilateral Primary open angle glaucoma or ocular hypertension
* Intra Ocular Pressure above 19 millimeters mercury at screening visit at 8:00 AM
* Stable visual field in last 6 months
* 6 weeks wash out from previous topical medications

Exclusion Criteria:

* Age

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Fornoni, Study Director — Alcon Research
Locations (1):
- Catania, Catania, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 patients suffering from POAG or ocular hypertension, with an intraocular pressure that was insufficiently controlled were recruited.
Pre-assignment Details: Subjects meeting the inclusion/exclusion criteria were enrolled.
Groups:
- Crossover Group ABB: Participants received Treatment A, which was concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.) for period 1 for 8 weeks. Then participants received Treatment B, which was fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.) for Period 2 (8 weeks) and Period 3 (8 weeks)
- Crossover Group BAA: Participants received Treatment B, which was fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.) for Period 1 (8 weeks). Then participants received Treatment A, which was concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.) for Period 2 (8 weeks) and Period 3 (8 weeks).
Period: First Intervention
Arm/Group | Crossover Group ABB | Crossover Group BAA
Started | 22 | 24
Completed | 18 | 20
Not Completed | 4 | 4
Period: Second Intervention
Arm/Group | Crossover Group ABB | Crossover Group BAA
Started | 18 | 20
Completed | 18 | 16
Not Completed | 0 | 4
Period: Third Intervention
Arm/Group | Crossover Group ABB | Crossover Group BAA
Started | 18 | 16
Completed | 17 | 14
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Population
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Intra Ocular Pressure (IOP)
Description: Intra Ocular Pressure, calculated as AUC (area under the curve) of IOP measured from 8.00 a.m. to 8.00 p.m, at different time-points
Time Frame: Baseline, end of each period (week 8, week 16, week 24)
Measure: Mean (Standard Deviation); unit: mm Hg (millimeters mercury)*week
Arm/Group | Crossover Group ABB | Crossover Group BAA
Number analyzed (Participants) | 22 | 24
mm Hg (millimeters mercury)*week
  Week 8 | 179.20 (25.42) | 191.89 (52.59)
  Week 16 | 188.82 (32.05) | 196.26 (59.07)
  Week 24 | 201.50 (41.01) | 191.93 (41.39)

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Treatment A: Participants received Treatment A, which was concomitant administration of travoprost 0.004% (ophthalmic drops, 1 drop/eye at approximately 19:45 p.m.) and brinzolamide 1% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.).
- Treatment B: Participants received Treatment B, which was fixed combination of timolol 0.5% and dorzolamide 2% (ophthalmic drops, 1 drop/eye, at 08:00 a.m. and at 20:00 p.m.), and travoprost vehicle (ophthalmic drops, 1 drop/eye, at approximately 19:45 p.m.).
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/24
Other Adverse Events (participants affected / at risk) | 11/22 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=22) | Treatment B (N=24)
Sternal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not drug related
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not drug related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=22) | Treatment B (N=24)
Conjunctivitis Allergic (Eye disorders) | 3 (3) | 1 (1)
Eye Irritation (Eye disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any formal presentation of data publication from this study has to be a joint presentation from both the Investigators and the Sponsor. Being the study multicentric, it is mandatory that the first publication is based on data from all the centres, analysed according to the protocol. Data from a single Centre can not be presented, unless there Is a formal agreement from the other Investigators and Alcon.